CLINICAL TRIAL: NCT02851329
Title: Association of Computed Tomography Phenotypic Signature With Progression-free Survival in Stage IV EGFR-mutant Non-small Cell Lung Cancer Undergoing Tyrosine Kinase Inhibitors
Brief Title: Therapeutic Resistance Prediction of Tyrosine Kinase Inhibitors
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Guangdong Academy of Medical Sciences (Other); West China Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chongwei Chi, Ph.D, Associate professor, Chinese Academy of Sciences
Other Study IDs: 20160728TRPN
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: stage IV EGFR-mutant; EGFR TKIs; progression-free survival; prognosis; computed tomography
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators propose a non-invasive prognostic tool for TKIs resistance in patients with stage IV EGFR-mutant non-small cell lung cancer (NSCLC) by computed tomography phenotypic features, which can be conveniently translated to facilitate the pre-therapy individualized management of EGFR TKIs in this disease.

DETAILED DESCRIPTION:
The investigators develop a multi-CT-phenotypic-feature-based classifier to predict TKI benefit and therapeutic resistance for stage IV EGFR-mutant non-small cell lung cancer (NSCLC). The investigators also compared its prognostic and predictive efficacy with single features and clinicopathological risk factors. An individualized nomogram integrated the classifier and three clinicopathological risk factors was built for clinical use. The prognostic accuracy of the proposed model was evaluated in two independent validation sets.

Nearly 500 patients will be enrolled in this clinical trial. Eligible patients were diagnosed with NSCLC, and stage IV according to the TNM system classification of the American Joint Committee on Cancer, presence of activating EGFR mutations, age 20 years or older, and no history of systemic anticancer therapy for advanced disease. Patients who underwent first-line or second-line EGFR TKIs were eligible for inclusion. All patients had to be capable of undergoing contrast-enhanced CT, and pretreatment CT was strictly controlled in two weeks before the EGFR TKIs starts. Patients who underwent resection for local advanced or metastatic disease were withdrawn from the study.

Therapeutic resistance was measured by PFS, as the time from the initiation of EGFR TKIs therapy to the date of confirmed disease progression or death. PFS was censored at the date of death from other causes, or the date of the last follow-up visit for progression-free patients.

The investigators will use extracted 1000 phenotypic features on the region of interest manually segmented by radiologists. The Lasso Cox regression model and Nomogram will be used to build a prognosis model for the therapeutic resistance prediction of EGFR TKIs for stage IV EGFR-mutant NSCLC. The Harrell's concordance index(C-index) of the proposed nomogram will be used to quantify the discrimination performance.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were diagnosed with NSCLC, and stage IV according to the TNM system classification of the American Joint Committee on Cancer.
* Presence of activating EGFR mutations.
* Age 20 years or older, and no history of systemic anticancer therapy for advanced disease.
* Patients who underwent first-line or second-line EGFR TKIs were eligible for inclusion.
* All patients had to be capable of undergoing contrast-enhanced CT, and pretreatment CT was strictly controlled in two weeks before the EGFR TKIs starts.

Exclusion Criteria:

* Based on the criteria above, patients who underwent resection for local advanced or metastatic disease were withdrawn from the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Currently, a cohort of 300 patients has already been collected from the collaborating hospitals. Next, the 3 hospitals will collect at least 200 patients within 1 years.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-03 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jiangdian Song, Ph.D., Principal Investigator — CAS Key Laboratory of Molecular Imaging, Institute of Automation, Chinese Academy of Sciences
Locations (1):
- Key Laboratory of Molecular Imaging, Chinese Academy of Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Crystal AS, Shaw AT, Sequist LV, Friboulet L, Niederst MJ, Lockerman EL, Frias RL, Gainor JF, Amzallag A, Greninger P, Lee D, Kalsy A, Gomez-Caraballo M, Elamine L, Howe E, Hur W, Lifshits E, Robinson HE, Katayama R, Faber AC, Awad MM, Ramaswamy S, Mino-Kenudson M, Iafrate AJ, Benes CH, Engelman JA. Patient-derived models of acquired resistance can identify effective drug combinations for cancer. Science. 2014 Dec 19;346(6216):1480-6. doi: 10.1126/science.1254721. Epub 2014 Nov 13. PMID 25394791
- [Background] Seto T, Kato T, Nishio M, Goto K, Atagi S, Hosomi Y, Yamamoto N, Hida T, Maemondo M, Nakagawa K, Nagase S, Okamoto I, Yamanaka T, Tajima K, Harada R, Fukuoka M, Yamamoto N. Erlotinib alone or with bevacizumab as first-line therapy in patients with advanced non-squamous non-small-cell lung cancer harbouring EGFR mutations (JO25567): an open-label, randomised, multicentre, phase 2 study. Lancet Oncol. 2014 Oct;15(11):1236-44. doi: 10.1016/S1470-2045(14)70381-X. Epub 2014 Aug 27. PMID 25175099
- [Background] Lambin P, van Stiphout RG, Starmans MH, Rios-Velazquez E, Nalbantov G, Aerts HJ, Roelofs E, van Elmpt W, Boutros PC, Granone P, Valentini V, Begg AC, De Ruysscher D, Dekker A. Predicting outcomes in radiation oncology--multifactorial decision support systems. Nat Rev Clin Oncol. 2013 Jan;10(1):27-40. doi: 10.1038/nrclinonc.2012.196. Epub 2012 Nov 20. PMID 23165123
- [Background] Balachandran VP, Gonen M, Smith JJ, DeMatteo RP. Nomograms in oncology: more than meets the eye. Lancet Oncol. 2015 Apr;16(4):e173-80. doi: 10.1016/S1470-2045(14)71116-7. PMID 25846097
- [Background] Miller VA, Hirsh V, Cadranel J, Chen YM, Park K, Kim SW, Zhou C, Su WC, Wang M, Sun Y, Heo DS, Crino L, Tan EH, Chao TY, Shahidi M, Cong XJ, Lorence RM, Yang JC. Afatinib versus placebo for patients with advanced, metastatic non-small-cell lung cancer after failure of erlotinib, gefitinib, or both, and one or two lines of chemotherapy (LUX-Lung 1): a phase 2b/3 randomised trial. Lancet Oncol. 2012 May;13(5):528-38. doi: 10.1016/S1470-2045(12)70087-6. Epub 2012 Mar 26. PMID 22452896